CLINICAL TRIAL: NCT07150143
Title: Comparative Effects of Connective Tissue Massage and Physical Modalities Added to Cervical and Scapulothoracic Stabilization Exercises on Pain, Function, and Endurance in Individuals With Chronic Neck Pain
Brief Title: Effects of Connective Tissue Massage and Physical Modalities Combined With Stabilization Exercises in Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, Assistant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-KAEK-63-22-07
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-specific Neck Pain
Keywords: non-specific neck pain; scapulothoracic stabilization exercises; connective tissue massage; electrotherapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Active Comparator): Each exercise session lasts 50 minutes, consisting of 10 minutes of warm-up, 30 minutes of stabilization exercises, and 10 minutes of cool-down. Stabilization exercises will be selected from an exercise pool according to the individual's needs, with progression ensured throughout the program. The exercises will be administered face-to-face twice a week for eight weeks, and participants will be provided with illustrated brochures and instructed to perform a one-hour home exercise program daily.
  Interventions: Other: Exercise
- Exercise, and Connective tissue massage (Experimental): Each exercise session lasts 50 minutes, consisting of 10 minutes of warm-up, 30 minutes of stabilization exercises, and 10 minutes of cool-down. Stabilization exercises will be selected from an exercise pool according to the individual's needs, with progression ensured throughout the program. The exercises will be administered face-to-face twice a week for eight weeks, and participants will be provided with illustrated brochures and instructed to perform a one-hour home exercise program daily. In this group, in addition to these exercises, connective tissue massage will be applied, starting from the basic regions and gradually incorporating other regions.
  Interventions: Other: Exercise; Other: Connective tissue massage
- Exercise, and Electro-physical modalities (Experimental): Each exercise session lasts 50 minutes, consisting of 10 minutes of warm-up, 30 minutes of stabilization exercises, and 10 minutes of cool-down. Stabilization exercises will be selected from an exercise pool according to the individual's needs, with progression ensured throughout the program. The exercises will be administered face-to-face twice a week for eight weeks, and participants will be provided with illustrated brochures and instructed to perform a one-hour home exercise program daily. Also, the electrotherapy program consists of 20 minutes of infrared therapy, continuous ultrasound will be applied to the right and left sides for 7 minutes each at an intensity of 2 W/cm², and 20 minutes of conventional TENS will be administered to the painful area.
  Interventions: Other: Exercise; Other: Infrared therapy; Other: Continuous ultrasound; Other: Conventional TENS

INTERVENTIONS:
Other: Exercise — Each exercise session lasts 50 minutes, consisting of a 10-minute warm-up, 30 minutes of stabilization exercises, and a 10-minute cool-down. Stabilization exercises are selected from an exercise pool according to the individual's needs, with progression ensuring throughout the program. The exercises will be administered face-to-face twice a week for eight weeks, and participants will be provided with illustrated brochures and instructed to perform a one-hour home exercise program daily.
Other: Connective tissue massage — Connective tissue massage will be applied, starting from the basic regions and gradually incorporating other regions.
  Arms: Exercise, and Connective tissue massage
Other: Infrared therapy — Infrared therapy will be applied for 20 minutes
  Arms: Exercise, and Electro-physical modalities
Other: Continuous ultrasound — Continuous ultrasound will be applied to the right and left sides for 7 minutes each at an intensity of 2 W/cm².
  Arms: Exercise, and Electro-physical modalities
Other: Conventional TENS — 20 minutes of conventional TENS will be administered to the painful area.
  Arms: Exercise, and Electro-physical modalities

SUMMARY:
This randomized, double-blinded controlled trial aims to investigate the comparative effects of connective tissue massage and physical modalities, when combined with cervical and scapulothoracic stabilization exercises, in individuals with chronic non-specific neck pain. A total of 51 participants aged 18-65 years will be randomly assigned into three groups. Group 1 will perform stabilization exercises alone, Group 2 will receive stabilization exercises plus connective tissue massage, and Group 3 will receive stabilization exercises plus electrotherapy modalities (infrared, continuous ultrasound, and TENS). The interventions will be conducted twice weekly for 8 weeks, and participants will also perform home-based exercises daily. Primary outcomes include pain, disability, and endurance, while secondary outcomes focus on quality of life, cervical range of motion, and scapular function.

DETAILED DESCRIPTION:
Chronic non-specific neck pain is a prevalent musculoskeletal disorder that adversely affects pain, functional capacity, and quality of life. Stabilization-based exercise programs are commonly recommended; however, the added benefits of connective tissue massage and physical modalities require further investigation.

This randomized, double-blinded controlled trial is designed to compare the effects of (1) stabilization exercises alone, (2) stabilization exercises combined with connective tissue massage, and (3) stabilization exercises combined with electrotherapy modalities (infrared therapy, continuous ultrasound, and TENS) on clinical outcomes in individuals with chronic non-specific neck pain.

A total of 51 participants between 18 and 65 years of age will be randomly allocated into three equal groups. All groups will receive supervised exercise sessions twice weekly for 8 weeks, each lasting 50 minutes (10 minutes of warm-up, 30 minutes of cervical and scapulothoracic stabilization, and 10 minutes of cool-down). Additionally, participants will be instructed to perform a one-hour home exercise program daily, supported with illustrated brochures.

The primary outcomes are:

* Pain (Bournemouth Neck Questionnaire)
* Disability (Neck Disability Index)
* Endurance (Deep Cervical Flexor Test)

The secondary outcomes are:

* Quality of life (WHOQOL-BREF)
* Cervical range of motion
* Scapular function (Lateral Scapular Slide Test and Scapular Dyskinesis Test)

By comparing these approaches, the study aims to determine whether the addition of connective tissue massage or physical modalities enhances the therapeutic effects of stabilization exercises on pain, function, and endurance in patients with chronic non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age,
* Having non-specific chronic neck pain localized to the posterior cervical spine between the occipital region and the spinous process of the first thoracic vertebra,
* Being able to cooperate with the assessments to be performed in the study.

Exclusion Criteria:

* Neck pain resulting from trauma within the past 6 months;
* A history of surgery related to cervical problems;
* Clinical signs of cervical radiculopathy and/or myelopathy;
* Inflammatory arthritis involving the cervical spine;
* Tumors or infections of the cervical spine;
* Vertebrobasilar artery insufficiency;
* Neurological disorders (such as multiple sclerosis, Parkinson's disease, or syringomyelia);
* Congenital anomalies affecting the spine; systemic diseases (such as diabetes mellitus);
* Shoulder pathologies (including tendinitis, bursitis, or capsulitis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | From enrollment to the end of treatment at 8 weeks
  To assess disability in neck pain, only the Neck Disability Index (NDI), which evaluates current pain and disability, was used. The NDI consists of 10 items grouped into 6 subdomains. Each item is scored on a scale from 0 to 5, with higher scores indicating greater levels of disability.
Deep Cervical Flexor Test | From enrollment to the end of treatment at 8 weeks.
  To evaluate deep neck flexor muscle endurance, the Deep Cervical Flexor Test was used. This test assesses the maximal contraction capacity of the deep cervical flexor muscles. It is performed in the supine position, with the participant lifting the head approximately 2.5 cm off the surface while maintaining chin retraction. The examiner places a hand under the participant's occiput. The test is terminated when cervical flexion is lost or the participant's head touches the examiner's hand, and the duration is recorded in seconds.
Cervical Range of Motion Assessment | From enrollment to the end of treatment at 8 weeks
  Cervical range of motion was assessed using a universal goniometer. The participant was seated in an upright position, and measurements were taken for cervical flexion, extension, right and left rotation, and right and left lateral flexion. For flexion and extension, the acromion was accepted as the pivot point, with the stationary arm held parallel to the ground and the movable arm aligned with the ear line. For rotation, a straight rod was placed between the participant's teeth, the midline of the head was accepted as the pivot point, the stationary arm was kept parallel to the ground, and the movable arm was aligned with the rod. For lateral flexion, the spinous process of C7 was accepted as the pivot point, the stationary arm was positioned parallel to the ground, and the movable arm was aligned with the spinous processes of the cervical vertebrae. Care was taken to ensure that the head was not rotated during the measurements.
Bournemouth Neck Questionnaire | From enrollment to the end of treatment at 8 weeks.
  For pain assessment, the Bournemouth Neck Questionnaire, which focuses on the participant's current symptoms over the past week, was used. The questionnaire evaluates aspects such as onset, localization, duration, type and characteristics of pain, aggravating and relieving factors, history of previous treatments, and accompanying symptoms. The Bournemouth Neck Questionnaire consists of 7 items, each scored on a scale from 0 to 10. The maximum score is 70, with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Quality of Life Assessment | From enrollment to the end of treatment at 8 weeks.
  The World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF) was used to assess the quality of life of the participants. The WHOQOL-BREF was developed by the World Health Organization and consists of six domains. Since each domain independently reflects the quality of life within its own scope, domain scores are calculated on a scale ranging from 4 to 20. Higher scores indicate better quality of life.
Lateral Scapular Slide Test | From enrollment to the end of treatment at 8 weeks.
  The Lateral Scapular Slide Test (LSST) is a clinical assessment used to evaluate scapular positioning and detect scapular dyskinesis by measuring the distance between the inferior angle of the scapula and the spinous process at various arm positions.
Scapular Dyskinesis Test | From enrollment to the end of treatment at 8 weeks.
  In the Scapular Dyskinesis Test, a load of 2.3 kg is used for individuals weighing 68.1 kg or more, and a load of 1.4 kg is used for those weighing less than 68.1 kg. Participants are instructed to hold the weights with the thumbs pointing upward, elbows extended, and shoulders in a neutral position, and to actively perform bilateral shoulder flexion and abduction. Each movement is repeated five times, during which scapular motion is observed. The presence of scapular winging or dysrhythmia during the movements is recorded as either "dyskinesis present" or "dyskinesis absent".
Scapular Retraction Test | From enrollment to the end of treatment at 8 weeks.
  The Scapular Retraction Test is used to grade the strength of the supraspinatus muscle. The test begins with the traditional Empty Can Test, in which the patient's shoulder is placed in internal rotation, 90 degrees of flexion, and the scapular plane position ("scaption"). The examiner applies a downward force to the patient's arm while the patient resists. The test is then repeated with the examiner manually stabilizing the scapula in a retracted position. To achieve this, the examiner's fingers firmly grasp the patient's anterior shoulder over the clavicle, while the forearm is positioned along the medial border of the scapula. The test is considered positive if rotator cuff strength is restored, as indicated by the patient's improved ability to resist the examiner's downward force compared with the traditional Empty Can Test.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu AKKURT, PhD, Study Director — Fenerbahçe University
Locations (1):
- Fenerbahçe Üniversitesi, Ataşehir, Istanbul, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT07150143/Prot_SAP_000.pdf